CLINICAL TRIAL: NCT06347159
Title: An Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of EDG-7500 in Adults With Hypertrophic Cardiomyopathy
Brief Title: A Study of EDG-7500 in Adults With Hypertrophic Cardiomyopathy (CIRRUS-HCM)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EDG-7500-102
Record Dates: First submitted 2024-03-18; First posted 2024-04-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-06

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: EDG-7500 Single Dose (Experimental)
  Interventions: Drug: EDG-7500
- Part B: EDG-7500 Multiple Dose in Adults with Obstructive Hypertrophic Cardiomyopathy (Experimental): EDG-7500 once daily for up to 28 days.
  Interventions: Drug: EDG-7500
- Part C: EDG-7500 Multiple Dose in Adults with Nonobstructive Hypertrophic Cardiomyopathy (Experimental): EDG-7500 once daily for up to 28 days.
  Interventions: Drug: EDG-7500
- Part D: EDG-7500 Multiple Dose in Adults with Hypertrophic Cardiomyopathy (Experimental): EDG-7500 daily for up to 18 months in new participants and participants who have completed Part B or C.
  Interventions: Drug: EDG-7500

INTERVENTIONS:
Drug: EDG-7500 — Liquid suspension formulation of EDG-7500
  Arms: Part A: EDG-7500 Single Dose
Drug: EDG-7500 — Solid oral formulation of EDG-7500
  Arms: Part B: EDG-7500 Multiple Dose in Adults with Obstructive Hypertrophic Cardiomyopathy; Part C: EDG-7500 Multiple Dose in Adults with Nonobstructive Hypertrophic Cardiomyopathy; Part D: EDG-7500 Multiple Dose in Adults with Hypertrophic Cardiomyopathy

SUMMARY:
This study is being conducted in order to understand the safety and effects of different doses of EDG-7500 as a single dose in adults with obstructive hypertrophic cardiomyopathy (oHCM) and as multiple doses in adults with obstructive or nonobstructive hypertrophic cardiomyopathy (nHCM).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or nonpregnant female, age ≥18 years to <85 years.
* Body mass index (BMI) ≥18 to <35 kg/m2; weight ≥50 kg at Screening (BMI ≥ 18 to < 40 kg/m2 is permitted for participants < 50 years).
* Diagnosed with hypertrophic cardiomyopathy at the time of Screening consistent with current American College of Cardiology Foundation/American Heart Association Guidelines.
* LVOT peak gradient ≥ 50 mmHg measured at rest or during the Valsalva maneuver as determined by echocardiography at Screening (Part A, B and D oHCM only).
* LVOT peak gradient < 30 mmHg measured at rest and < 50 mmHg measured during the Valsalva maneuver as determined by echocardiography at Screening (Part C and D nHCM only).
* Documented left ventricular ejection fraction (LVEF) ≥ 0.60 at Screening.
* New York Heart Association (NYHA) Classification II-III at Screening.
* Kansas City Cardiomyopathy Questionnaire-Clinical Summary Score (KCCQ-CSS) < 85 at Screening.
* NT-proBNP ≥ 300 pg/mL (NT-proBNP ≥ 225 pg/mL is permitted for African American participants) (Part C and D nHCM only).

Key Exclusion Criteria:

* Invasive septal reduction therapy < 180 days prior to or during Screening.
* Documented history of active or untreated obstructive coronary artery disease during Screening or treated for obstructive coronary artery disease < 180 days prior to Screening.
* Documented history of myocardial infarction with residual wall motion abnormalities < 180 days prior to or during Screening.
* Significant valvular heart disease (moderate or greater aortic stenosis or regurgitation, moderate or greater mitral stenosis or regurgitation not due to systolic anterior motion of the mitral valve)
* History of LV systolic dysfunction (LVEF < 0.45) or stress cardiomyopathy at any time.
* Known or suspected infiltrative or storage disorder causing cardiac hypertrophy that may mimic HCM, such as Fabry disease, amyloidosis, or Noonan syndrome with LV hypertrophy.
* A history of unexplained syncope <180 days prior to or during Screening.
* A history of sustained ventricular tachyarrhythmia or sudden cardiac arrest < 180 days prior or during Screening.
* A history of known appropriate implantable cardioverter defibrillator (ICD) discharge <180 days prior to or during Screening or ICD implanted < 14 days prior to Screening.
* History of permanent AF or atrial flutter. Documented AF or atrial flutter requiring rhythm restoring treatment < 180 days prior to Screening Visit (participants with documented AF or atrial flutter requiring rhythm restoring treatment ≥ 180 days prior to Screening require adequate anticoagulation.)
* Fridericia-corrected QT interval (QTcF) ≥480 ms or any other ECG abnormality considered by the Investigator or Medical Monitor to pose a risk to participant safety at Screening (QTcF < 530 ms is permitted for participants with documented bundle branch blockage (BBB) and/or cardiac pacing).
* Receiving a CMI (e.g., Camzyos® [mavacamten] or aficamten) < 90 days prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | From screening through study completion (Part A: Up to 38 days; Part B and C: Up to 73 days; Part D: Up to 18 months)

SECONDARY OUTCOMES:
Change from baseline in left ventricular outflow tract (LVOT) gradient | From baseline through study completion (Part A: Up to 10 days; Part B: Up to 38 days; Part D: Up to 18 months)
  Resting and post-Valsalva LVOT gradient by echocardiography
Pharmacokinetic parameters of EDG-7500 as measured by maximum plasma concentration (Cmax) | From baseline through study completion (Part A: Up to 10 days)
Change from baseline in cardiac biomarkers | From baseline through study completion (Part B and C: Up to 38 days; Part D: Up to 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Edgewise Therapeutics, Inc.
Locations (20):
- United States (20):
  - University of California, San Francisco, San Francisco, California
  - Stanford University Hospital / Stanford Health Care, Stanford, California
  - Emory Clinic, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Michigan Medicine - Michigan Clinical Research Unit, Ann Arbor, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Morristown Medical Center (Atlantic Health System), Morristown, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Health Medical Center - HCM Program Office (Study open to existing NYU patients only), New York, New York
  - Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - Duke Health Center Arringdon, Morrisville, North Carolina
  - The Lindner Research Center at Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Hospital of the University of Pennsylvania (University of Pennsylvania School of Medicine), Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Virginia Heart and Vascular Center Fontaine, Charlottesville, Virginia
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No